CLINICAL TRIAL: NCT03768895
Title: Assement of the Morphological Characteristics of the Hips and Correlating Them With the Pathology Found
Status: Completed | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Maria Pilar López Royo, Principal Investigator, Universidad de Zaragoza
Other Study IDs: MRI center
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Hip Pain Chronic; Musculoskeletal Disease; Femoral Anteversion
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI group: The criteria for patient inclusion were: Age > 18 years old, who had realised a pelvis MRI for any cause at MRI Center. Exclusion criteria included age < 18 years old, inadequate imaging quality, medical history likely to affect pelvic and hip morphometry: pelvic oncological disease, infection or inflammatory arthritis, postsurgical change disruptions, soft tissue abnormality, avascular necrosis, or pelvic and hip fracture.
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — The technique used was coronal and axial T1 and T2*WI sequences of the pelvis and femurs.
  The MRI machine used is a HITACHI AIRIS-II1 model, with permanent vertical magnetic field of 0.3 Tesla, and the used sequences areT1, T2*WI.

SUMMARY:
The investigators' objective is the anatomical analysis of hips studied through MRI, assessing their morphological characteristics and correlating them with the pathology found.

A retrospective search was performed using a database of consecutive reports of 137 adults pelvis MRI examinations obtained at MRI center in Zaragoza.

In all the images the investigators are going to measure the ischiofemoral space, quadratus femoris space, cervicodiaphysal angle and femoral version angle. The investigators evaluated different qualitative changes in the signal intensity of the quadratus femoris muscle as normal, edema, fatty infiltration or atrophy, and of the gluteus muscles as tendinopathy or atrophy, too.

DETAILED DESCRIPTION:
The investigators' objective is the anatomical analysis of hips studied through MRI, assessing their morphological characteristics and correlating them with the pathology found.

A retrospective search was performed using a database of consecutive reports of 137 adults pelvis MRI examinations obtained at MRI center in Zaragoza.

The investigators create a protocol for a retrospective review study, with the aim of analysis all the recorded MRI findings during this time. The criteria for patient inclusion were: Age > 18 years old, who had realised a pelvis MRI for any cause at MRI Center. Exclusion criteria included age < 18 years old, inadequate imaging quality, medical history likely to affect pelvic and hip morphometry: pelvic oncological disease, infection or inflammatory arthritis, postsurgical change disruptions, soft tissue abnormality, avascular necrosis, or pelvic and hip fracture.

In all the images the investigators are going to measure the ischiofemoral space, quadratus femoris space, cervicodiaphysal angle and femoral version angle. The investigators evaluated different qualitative changes in the signal intensity of the quadratus femoris muscle as normal, edema, fatty infiltration or atrophy, and of the gluteus muscles as tendinopathy or atrophy, too.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old

Exclusion Criteria:

* Age < 18 years old
* Inadequate imaging quality
* Medical history likely to affect pelvic and hip morphometry: pelvic oncological disease, infection or inflammatory arthritis, postsurgical change disruptions, soft tissue abnormality, avascular necrosis, or pelvic and hip fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who had realised a pelvis MRI for any cause at MRI Center in Zaragoza.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Ischiofemoral Space | 1 day
  the smallest distance between the lateral cortex of the ischial tuberosity and medial cortex of the lesser trochanter.
Quadratus Femoris Space | 1 day
  the smallest space for passage of the quadratus femoris muscle delimited by the superolateral surface of the hamstring tendons and the posteromedial surface of the iliopsoas tendón or lesser trochanter.
Cervicodiaphyseal angle | 1 day
  The cervicodiaphyseal angle is formed by the axis of the femoral neck that joins the femoral head with the axis of the femoral shaft.
Femoral version | 1 day
  The femoral version or femoral torsion angle is called the projection on the transverse plane of a longitudinal axis of the femoral neck at the center of the femoral head

CONTACTS AND LOCATIONS:
Locations (1):
- Dra. Roca Diagnóstico Médico. CEMEDI, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided